CLINICAL TRIAL: NCT06229041
Title: Total Neoadjuvant Treatment ±Immunotherapy for High Risk Locally Advanced Rectal Cancer (TNTi)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Beijing Nanjiao Cancer Hospital (Unknown)
Responsible Party: Principal Investigator, Aiwen Wu, Chief of Gastrointestinal Center Unit III, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUCH R07
Record Dates: First submitted 2024-01-09; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; High risk; Immunotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Neoadjuvant Treatment ＋Immunotherapy (Experimental)
  Interventions: Drug: Camrelizumab ＋Immunotherapy
- Total Neoadjuvant Treatment (No Intervention)

INTERVENTIONS:
Drug: Camrelizumab ＋Immunotherapy — Camrelizumab was used in preoperative treatment.
  Arms: Total Neoadjuvant Treatment ＋Immunotherapy

SUMMARY:
The goal of this clinical trial is to compare the PCR rate between Total Neoadjuvant Treatment ±Immunotherapy in high risk locally advanced rectal cancer. The main questions it aims to answer are:

* The PCR rate between the two groups
* The 3years DFS between the two groups
* Chemoradiotherapy and immunotherapy toxicity
* Postoperative complications Participants will receive total neoadjuvant treatment ±immunotherapy followed by surgery.

Researchers will compare neoadjuvant treatment ±immunotherapy to see the PCR rate.

ELIGIBILITY:
Inclusion Criteria:

1. >18，<75 years old
2. ECOG score 0-1
3. colorectal adenocarcinoma confirmed by pathology
4. The distance between the lower margin of the tumor and the anal margin is ≤12cm or the distance between the anorectal ring (ARJ) is ≤8cm
5. The initial local MRI stage was T4b, or mrN2, or positive MRF, or positive EMVI, or lateral lymph node metastasis (mrLLND+)
6. No evidence of distant metastasis
7. No history of pelvic radiotherapy
8. No history of rectal cancer surgery or chemotherapy
9. Systemic infections that do not require antibiotic treatment
10. Not associated with immune system diseases
11. Blood routine: ANC>1.5 cells/mm3, HGB>9.0g /dL, PLT>800,000/mm3
12. Blood biochemistry: total bilirubin ≤1.5xULN, AST≤2.5xULN, ALT≤2.5xULN;
13. Serum creatinine ≤1.5 times the upper limit of normal and endogenous creatinine clearance ≥50mL/min (Cockcroft-Gault formula)
14. Patients with well-controlled hypertension were allowed to be enrolled
15. International Standardized ratio (INR), activated partial thromboplastin time (aPTT) ≤1.5 times the upper limit of normal value (only applicable to patients who have not received anticoagulant therapy; Patients receiving anticoagulant therapy should keep anticoagulants within the therapeutic requirements)
16. Normal or abnormal FT3, FT4 and TSH have no clinical significance
17. Normal cardiac function, that is, normal or abnormal ECG examination has no clinical significance, and left ventricular ejection fraction (LVEF) shown by cardiac ultrasound is greater than 50%
18. The patient read and signed the informed consent of this study and agreed to participate in this study
19. The subjects voluntarily joined the study, signed the informed consent, had good compliance and cooperated with the follow-up. It is recommended that all patients provide tumor tissue samples (preferably fresh) for pathological/genetic testing prior to enrollment
20. Fertile men or women with the possibility of becoming pregnant must use a highly effective contraceptive method throughout the trial and continue contraception for 12 months after the end of treatment

Exclusion Criteria:

1. Recurrent rectal cancer
2. Microsatellite instability (MSI) or mismatch repair gene deletion (dMMR)
3. The patient has had other malignancies in the past 5 years (in addition to properly treated basal cell carcinoma and skin squamous cell carcinoma)
4. The patient has had arterial embolic diseases in the past 6 months, such as angina pectoris, MI, TIA, CVA, etc.
5. Have received other types of anti-tumor or experimental therapy
6. The patient is a pregnant or lactating woman
7. The patient has other diseases or mental disorders that may affect the patient's participation in this study
8. Patients who have previously received anti-PD-1, anti-PD-L1, anti-PD-L2 therapy or VEGFR TKI therapy.
9. Major surgical procedures were performed/received within 4 weeks prior to the first administration of the study drug or the side effects of which have not yet recovered, live vaccination, immunotherapy, and radiotherapy within 2 weeks.
10. Study patients who had received hematopoietic stimulating factors, such as granulocyte colony-stimulating factor (G-CSF), erythropoietin, etc., within 1 week before the first administration of the drug.
11. Known allergy to the investigational drug and its components
12. Active lung disease (interstitial pneumonia, pneumonia, obstructive pulmonary disease, asthma) or a history of active tuberculosis.
13. Have any clinical problems beyond your control, including but not limited to:

    a persistent or active (severe) infection b Poorly controlled hypertension (persistent blood pressure greater than 150/90 MMHG) c Poorly controlled diabetes mellitus d Heart disease (Grade III/IV congestive heart failure or heart block as defined by the Heart Society of New York) e Have or suspect an autoimmune disease, or a history of autoimmune disease or syndromes requiring treatment with a steroid/immunosuppressive system, such as hypophysitis, colitis, hepatitis, nephritis, hyperthyroidism, hypothyroidism, etc.;
14. Other severe, acute, or chronic medical conditions or abnormalities in laboratory tests that the investigator determines may increase the risk associated with study participation or may interfere with the interpretation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
The PCR rate between total neoadjuvant treatment ±immunotherapy | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No